CLINICAL TRIAL: NCT05068193
Title: A Randomized, Open-label, Single Dose, Two-way Crossover Study to Compare the Pharmacokinetics and Bioequivalence of "BR2008" With "BR2008-1" in Healthy Volunteers
Brief Title: A Clinical Trial to Compare the Pharmacokinetics and Bioequivalence of "BR2008" With "BR2008-1" in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-RGR-CT-101
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2021-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Other): The investigational products will be administered according to the treatment groups(BR2008, BR2008-1) assigned to each sequence group in Period I and Period II.
  *Sequence 1
  [Period I] Administration of BR2008-1 (single dose)
  - Wash out for 2 weeks
  [Period II] Administration of BR2008 (single dose)
  Interventions: Drug: BR2008-1 (R); Drug: BR2008 (T)
- Sequence 2 (Other): The investigational products will be administered according to the treatment groups(BR2008, BR2008-1) assigned to each sequence group in Period I and Period II.
  *Sequence 2
  [Period I] Administration of BR2008 (single dose)
  * Wash out for 2 weeks
  [Period II] Administration of BR2008-1 (single dose)
  Interventions: Drug: BR2008-1 (R); Drug: BR2008 (T)

INTERVENTIONS:
Drug: BR2008-1 (R) — After fasting at least 10 hours, two tablets of BR2008-1 will be administered orally with 150mL of water around 8 a.m.
Drug: BR2008 (T) — After fasting at least 10 hours, one tablet of BR2008 will be administered orally with 150mL of water around 8 a.m.

SUMMARY:
A clinical trial to compare the pharmacokinetics and bioequivalence of BR2008 with BR2008-1 in healthy volunteers

ELIGIBILITY:
<Inclusion Criteria>

1. Healthy adults aged over 19 years at screening
2. Those who have no congenital or chronic diseases and have no abnormal symptoms or findings based on medical examination results
3. Determined to be eligible subjects as a result of clinical laboratory tests and electrocardiography performed according to this protocol at screening
4. Those who have calculated body mass index(BMI) within the range of 18.0 to 30.0 kg/m2
5. Those who do not have a history of the psychiatric diseases within the last 5 years before screening
6. Those who do not have a history of gastrointestinal diseases (e.g., Crohn's disease, ulcer, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (however, simple appendectomy or hernia repair are excluded) that may affect the absorption of drugs
7. Voluntarily decide to participate in the study and provide written consent to follow the study directions after listening to and fully understanding the detailed explanation on this study

<Exclusion Criteria>

1. Those who took drugs inducing and inhibiting drug-metabolizing enzymes, such as barbital, within 30 days prior to the first administration date, or took any drugs that may the clinical trial
2. Those who continue to drink alcohol (Male: >5 units/week, Female: >2.5 units/week) within 1 month prior to the first administration date
3. Those who continue to smoke (>10 cigarettes/day) or cannot stop smoking during hospitalization throughout the entire period from the date of 48 hours before the first administration of the investigational product to the last pharmacokinetic blood sampling
4. Those who have been determined by the investigator to be ineligible to participate in the clinical trial
5. Those who have participated in another clinical trial or bioequivalence test (the last day of administration of the investigational product or bioequivalence test drug) within 6 months prior to the first administration date
6. Those who have donated whole blood within 2 months, or donated blood components (apheresis) within 2 weeks, or who have received a blood transfusion within 30 days prior to screening
7. Those who do not agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy using a medically acceptable methods of contraception throughout the entire period from the date of the first administration of the investigational product to 8 weeks after the last administration of the investigational product
8. Those with severe hepatic impairment, or any of the following results in the screening tests

   * Total bilirubin ≥ 1.5 x ULN
   * AST(SGOT) or ALT(SGPT) ≥ 2 x ULN
   * r-GTP ≥ 1.5 x ULN
9. Those with severe renal impairment, or serum creatinine levels upper than 1.5 times of ULN
10. Those with a predisposition to bleeding, or taking anticoagulants(Warfarin, phenprocoumon), or taking concomitant medications that increase the risk of bleeding
11. Those with cardiovascular disease (heart ischemia and infarction)
12. Those with systolic blood pressure<90mmHg or >140mmHg, or diastolic blood pressure <60mmHg or >90mmHg
13. Those who have hypersensitivity reactions to "BR2008" or "BR2008-1"
14. Pregnant woman, potentially pregnant woman, or breast-feeding woman

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
AUCt | 0-120 hours after administration
  Area under the plasma drug concentration-time curve from time 0 to time t of BR2008 and BR2008-1
Cmax | 0-120 hours after administration
  Maximum concentration of drug in plasma of BR2008 and BR2008-1

CONTACTS AND LOCATIONS:
Locations (1):
- Bestian Hospital, Osŏng, South Korea